CLINICAL TRIAL: NCT00126698
Title: Use of Antibiotic Prophylaxis on Urethral Catheter Withdrawal: A Randomized Double-Blind Placebo-Controlled Trial
Brief Title: Prophylactic Antibiotics on Urethral Catheter Withdrawal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2005-01; CAD-Trial
Record Dates: First submitted 2005-08-02; First posted 2005-08-04 (Estimated); Last update posted 2007-04-19 (Estimated); Status verified 2007-04

CONDITIONS: Urinary Tract Infection; Bacteriuria
Keywords: Bacteriuria; Urinary Catheter; Urinary tract infection; Prophylaxis; Urinary catheter removal
MeSH Terms: conditions — Urinary Tract Infections; Bacteriuria | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Ciprofloxacin

INTERVENTIONS:
Drug: trimethoprim-sulfamethoxazole
Drug: ciprofloxacin

SUMMARY:
Urinary-tract infection (UTI) is the most common type of hospital-acquired infection (30% of all). The purpose of this study is to determine whether antibiotic prophylaxis for urinary catheter removal is useful at preventing catheter-associated urinary-tract infection.

DETAILED DESCRIPTION:
Urinary-tract infection (UTI) is the most common type of hospital-acquired infection (30% of all). The researchers undertake a double-blind, placebo-controlled trial to assess the efficacy of single-dose therapy of trimethoprim-sulfamethoxazole or ciprofloxacin, versus placebo therapy in selected groups of surgical patients who had bladder drainage scheduled to last longer than 3 days.

ELIGIBILITY:
Inclusion Criteria:

* Urethral catheter in situ for at least 3 days (72h)

Exclusion Criteria:

* Pregnancy
* Impaired renal or hepatic function (serum creatinine > 150 mmol/l, serum transaminases > 75 IU/l)
* Fever
* Symptomatic urinary tract infection
* Antibiotic use ≤ 48 hours before urinary catheter removal
* Allergy to trimethoprim-sulfamethoxazole or ciprofloxacin
* Urologic pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Symptomatic bacteriuria
Asymptomatic bacteriuria

SECONDARY OUTCOMES:
Antibiotic resistance patterns

CONTACTS AND LOCATIONS:
Overall Officials: M. Tersmette, MD, PhD, Study Director — Sint Antonius Hospital, Nieuwegein
Locations (1):
- Sint Antonius Hospital, Nieuwegein, Utrecht, Netherlands